CLINICAL TRIAL: NCT05789381
Title: Patient Satisfaction and Abbreviated Postpartum Magnesium Sulfate for Preeclampsia With Severe Features: a Randomized Controlled Trial
Brief Title: Patient Satisfaction With Abbreviated Postpartum Magnesium Sulfate for Severe Preeclampsia
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Feasibility reassessed, study design reevaluated, project withdrawn
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB22-0450
Record Dates: First submitted 2023-03-01; First posted 2023-03-29 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-10

CONDITIONS: Patient Satisfaction
Keywords: preeclampsia; pregnancy; postpartum; magnesium; satisfaction; breastfeeding
MeSH Terms: conditions — Patient Satisfaction; Pre-Eclampsia; Personal Satisfaction; Breast Feeding | interventions — Magnesium Sulfate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 24 hours postpartum magnesium sulfate (Active Comparator)
  Interventions: Procedure: Magnesium sulfate
- 12 hours postpartum magnesium sulfate (Experimental)
  Interventions: Procedure: Magnesium sulfate

INTERVENTIONS:
Procedure: Magnesium sulfate — This drug is commonly used on labor and delivery and in the postpartum period and is easily ordered through the electronic medical record and provided. This drug requires no specific storage for research study purposes as the drug is already being administered per standard of care and national and international guidelines. The only change is in the duration of therapy. This is NOT considered an off label use of the drug and does not require any form of exemption determination. Magnesium for severe preeclampsia is often given for anywhere from 12 to 24 hours postpartum depending on the clinical scenario, provider preference, and patient symptoms/adverse reactions to the medication.

SUMMARY:
Preeclampsia is a common and potentially devastating disease that affects only pregnant or postpartum patients. It is a leading cause of maternal mortality not only worldwide, but in the United States as well. As the medical field has advanced in many regards, including improved treatment for prevention of severe preeclampsia or even eclamptic seizures, the strain on pregnant and postpartum people has remained relatively unchanged. The most successful and widely used management of severe preeclampsia is magnesium sulfate, an intravenous infusion used to help prevent eclamptic seizures which can be additionally life threatening. While magnesium can be efficacious, it comes with some hindrances. Notably, magnesium itself can make patients feel ill-weak, confused, lethargic, "foggy", and even somnolent in cases of toxicity. Other adverse effects include pulmonary edema, and cardiac arrhythmias or even coma. These effects are common and concerning enough that it is regular practice to examine patients at the bedside with a full neurological exam every 2 hours while they are on magnesium, which is typically a course of at least 24 hours straight. Additionally, patients typically have a foley catheter in place to monitor urine output as magnesium can cause kidney injury, and they are bedbound because of the lethargy and concern for falls. In the postpartum period this has significant negative impacts on patients bonding with their newborn, initiating breast or chest feeding, walking, voiding, and aiding in faster postpartum recovery. While the implications of a life threatening medical diagnosis are devastating for many patients, the trauma that can be caused by being away from a patient's newborn or not feeling in control of the patients own body postpartum are issues that are finally starting to be recognized. While magnesium is necessary, there may be ways to treat patients while maintaining independence, mental health and sense of selves especially in the sensitive postpartum period. The investigators hypothesis is that, in a carefully selected group of patients with severe preeclampsia, 12 hours of magnesium sulfate leads to improved patient satisfaction, increased breastfeeding postpartum, as well as other markers of enhanced postpartum recovery, and lack of worsening symptoms or persistently elevated blood pressure in comparison to 24 hours of magnesium.

DETAILED DESCRIPTION:
1. Visit 1: the screening, consent and randomization visit. This takes place in the Family Birth Center as described above. The patient is approached for consent, randomized, and receives the study intervention in the postpartum period. Randomization will be performed through REDCap using permuted block technique. A permuted block randomization procedure will be used to formulate assignment lists in order to assure close to equal numbers of subjects in each treatment group. A uniform block size of 4 will be used, and the allocation ratio within each unit will be 1. A list of random digits (0-9) will be generated by a computer based random number generator. The list will then be transformed into a randomization schedule. Using a block size of four subjects, with four potential treatment groups, a permutation block assignment list will be created. Because of the block size, an allocation ratio of 1 will be assured after each subsequent group of eight subjects is allocated. Randomization will be performed using a computer-generated sequence in two blocks. Sequentially numbered opaque envelopes displaying only the randomization number on the outside will then be used. These envelopes will be stored in a locked closet on the labor and delivery unit.

   Blinding: Given the nature of the study, neither patients nor the covering provider can be blinded.

   Prior to discharge, patients receive the WOMB postnatal satisfaction questionnaire (WOMBPNSQ) and this is all considered the same visit (the labor and delivery visit).
2. Visit 2: this refers to the Postpartum visit. At anywhere from 2 to 12 weeks postpartum, the patient will come to see their provider for follow up care. At this visit, it is standard of care to collect the EDPS depression survey. This score will be collected for study data from the electronic medical record.

Patients will be approached if they have a diagnosis of preeclampsia with severe features. Patients who consent to participate in the study and are eligible will be randomized into 24 hours of magnesium therapy or 12 hours of magnesium therapy in the postpartum period. Magnesium levels will be obtained if indicated by standard protocol by patient symptoms and will be defined as magnesium level greater than 8.4 mg/dL or symptoms such as hyporeflexia, pulmonary edema, altered mental status. Patients will be asked to complete two surveys in the postpartum period, one for depression scoring and one for patient satisfaction in the postpartum period. The patient satisfaction survey will be administered prior to discharge from the hospital postpartum. The depression score survey will be administered at the patient's postpartum visit, as is the standard of care at all postpartum visits regardless of medical diagnoses.

Progression of symptoms/presence of symptoms is something that is subjectively measured by the physician team when rounding on the patient, by the nurses when assessing the patient, and is clearly documented in progress notes throughout the day and the patient's inpatient admission. Blood pressures are documented in the chart at regular intervals when they are recorded on the floor, and are easily accessed in the Vitals section of the EMR. The investigators outcome measure is not "improved" breastfeeding, but breastfeeding as a binomial variable (yes/no) and this is also clearly documented in the chart in progress note from the physician team, nursing team, and lactation team. This measure is regularly recorded within the investigators department for data collection for the entire Family Birthing Center. I have previously deleted maternal-neonatal bonding as an outcome measure, this is no longer a measure in investigators study. Magnesium toxicity is first suspected clinically and would be documented in the progress note section of the EMR, and it is confirmed with serum measurement of magnesium level (>8.4). This is documented in the Results Review/Laboratory section of the EMR and is easily accessible in the chart. Patient/maternal satisfaction with birth experience and postnatal experience will be evaluated by the WOMBPNSQ survey and postpartum depression will be evaluated by the Edinburgh survey.

Foley catheter removal is documented by nursing in the intake/output section of the medical record. Time to ambulation will be extrapolated by rounding notes from the care team.

Continuation/discontinuation rules: if the patient is randomized to the 12 hour magnesium arm and has worsening labs, uncontrollable blood pressures, or worsening headache/neurologic symptoms, they are deemed at a higher risk of eclamptic seizure and will therefore receive a full 24 hours of magnesium as is the standard of medical care. They will remain enrolled in the study, not be withdrawn, and be analyzed by intention to treat as they were randomized to the 12 hour arm. If the patient is randomized to the 24 hour arm, they will continue until 24 hours unless they have signs/symptoms of magnesium toxicity or if they self-withdraw from the study arm.

Length of study: For the individual patient, involvement in the study will last from enrollment until the postpartum appointment, which may be as far out as 10-12 weeks postpartum. Access to the patient's chart and information for the purposes of data extraction and analysis and completion of the study, manuscript preparation and submission, will last up to 3 years. The investigators will continue to store this information for 3 years before destroying all data collected.

ELIGIBILITY:
Inclusion Criteria:

* • Pregnancy >20 weeks EGA

  * Age 18 to 50
  * English speaking
  * Pre-eclampsia or superimposed pre-eclampsia with severe features diagnosed prior to delivery (antepartum), during labor and delivery (intrapartum)
  * Diagnosis of preeclampsia with severe features diagnosed undergoing induction of labor, spontaneous labor, or cesarean delivery (scheduled or unscheduled) delivering at the University of Chicago Family Birth Center
  * *Pre-eclampsia: is defined as new onset hypertension in pregnancy after 20 weeks gestation with proteinuria.
  * Pre-eclampsia with severe features may occur with or without proteinuria if ANY one of the following "severe features" are diagnosed: blood pressure >160/>110 sustained over 2 values 15 minutes apart, creatinine >1.1 or double patient baseline, liver function tests/AST and ALT double the upper limit of normal, persistent headache despite medication, pulmonary edema, right upper quadrant pain, platelet count <100,000.

Exclusion Criteria:

* • AKI or h/o CKD ( Cr >1.1)

  * HELLP syndrome (LFT's twice the upper limit of normal or platelets <100 not secondary to gestational or idiopathic thrombocytopenia with evidence of hemolysis by LDH levels or schistocytes on blood smear).
  * Eclampsia
  * Uncontrollable blood pressures requiring higher level of care such as in the intensive care unit
  * Diuresis < 30cc/kg /hr
  * Patients with neurologic signs or symptoms such as headache that does not remit with medication, blurred vision
  * Patients with ongoing right upper quadrant pain as a symptom of pre-eclampsia
  * Patients with other contraindications to magnesium prophylaxis such as myasthenia gravis, pulmonary edema

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
Patient satisfaction | Up until hospital discharge (assessed up until day 7)
  Patient satisfaction will be measured using the WOMB postnatal satisfaction questionnaire (WOMBPNSQ) which is a standardized survey instrument for postpartum patient satisfaction. This survey instrument has multiple versions with the most recent version consisting of 39 questions, measured on a Likert scale with answers ranging from 1 (least) to 7 (most). The higher scores will mean a better outcome or better patient satisfaction.

SECONDARY OUTCOMES:
Breastfeeding initiation | Up until 12 weeks postpartum
  Measured by patients report of "yes" or "no".
Magnesium toxicity | Up until 3 days postpartum
  Magnesium toxicity will be measured with the following possible criteria: lab values (magnesium >8.4 mg/dL) or symptoms (lethargy, altered mental status, hyporeflexia, pulmonary edema).
Worsening preeclampsia | Up until 7 days postpartum
  Worsening preeclampsia will be measured as clinical findings such as persistent headache, vision changes and right upper quadrant pain by postpartum day #3 and postpartum day #7. Measured by number of participants with elevated blood pressures recorded through the remote monitoring system and/or at their postpartum visits.
Persistently elevated blood pressure | Up until 7 days postpartum
  Persistently elevated blood pressure will be monitored by a home blood pressure cuff which is given to patients prior to hospital discharge when they have a diagnosis of preeclampsia. The home monitoring system is linked to a phone app which is already in use by the University of Chicago and triggers an alert when blood pressures are above 160 systolic or 110 diastolic. With a severe range blood pressure as described, an assessment by the physician on call is prompted. Persistently elevated blood pressures could also be mild range, meaning 140-159 systolic or 90-109 diastolic, and could prompt initiation of antihypertensive medication and would be included in outcomes measured for persistently elevated blood pressure.
Need for antihypertensive medication after discharge | Up until 12 weeks postpartum
  The decision to begin antihypertensive medication after discharge is closely linked to persistently elevated blood pressures, which is up to the discretion of the managing physician, but would be given if there were persistently elevated blood pressures in the severe range, 160 systolic or 110 diastolic. Medication is often also initiated when blood pressures are persistently in the mild range (140-159 systolic or 90-109 diastolic), meaning that >50% of measured blood pressure are within these ranges.
Maternal complications | Up until 12 weeks postpartum
  Pulmonary edema, seizure, ICU admission
Postpartum length of stay | Up until hospital discharge (assessed up until day 7)
  Measured in days
Postpartum depression | Up until 12 weeks postpartum
  The assessment of postpartum depression is a standard component of postpartum care. At the participant's postpartum visit they will be administered the Edinburgh Postnatal Depression Scale survey (EPDS). This consists of 10 questions, with a maximum score of 30. Possible depression is considered a score higher than 10. Questions 1, 2 and 4 are scored as 0, 1, 2, 3 and questions 3, 5, and 10 are reverse scored, with the top box scored as a 3 and the bottom box scored as 0. The final question asks about suicidal thoughts and always prompts further evaluation and assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Joana Lopes Perdigao, MD, Principal Investigator — University of Chicago

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bell MJ. A historical overview of preeclampsia-eclampsia. J Obstet Gynecol Neonatal Nurs. 2010 Sep-Oct;39(5):510-8. doi: 10.1111/j.1552-6909.2010.01172.x. PMID 20919997
- [Background] Alexander JM, McIntire DD, Leveno KJ, Cunningham FG. Selective magnesium sulfate prophylaxis for the prevention of eclampsia in women with gestational hypertension. Obstet Gynecol. 2006 Oct;108(4):826-32. doi: 10.1097/01.AOG.0000235721.88349.80. PMID 17012442
- [Background] Witlin AG, Sibai BM. Magnesium sulfate therapy in preeclampsia and eclampsia. Obstet Gynecol. 1998 Nov;92(5):883-9. doi: 10.1016/s0029-7844(98)00277-4. PMID 9794688
- [Background] Sibai BM. Magnesium sulfate prophylaxis in preeclampsia: Lessons learned from recent trials. Am J Obstet Gynecol. 2004 Jun;190(6):1520-6. doi: 10.1016/j.ajog.2003.12.057. PMID 15284724
- [Background] Fontenot MT, Lewis DF, Frederick JB, Wang Y, DeFranco EA, Groome LJ, Evans AT. A prospective randomized trial of magnesium sulfate in severe preeclampsia: use of diuresis as a clinical parameter to determine the duration of postpartum therapy. Am J Obstet Gynecol. 2005 Jun;192(6):1788-93; discussion 1793-4. doi: 10.1016/j.ajog.2004.12.056. PMID 15970809
- [Background] Vigil-De Gracia P, Ramirez R, Duran Y, Quintero A. Magnesium sulfate for 6 vs 24 hours post delivery in patients who received magnesium sulfate for less than 8 hours before birth: a randomized clinical trial. BMC Pregnancy Childbirth. 2017 Jul 24;17(1):241. doi: 10.1186/s12884-017-1424-3. PMID 28738788
- [Background] Altman D, Carroli G, Duley L, Farrell B, Moodley J, Neilson J, Smith D; Magpie Trial Collaboration Group. Do women with pre-eclampsia, and their babies, benefit from magnesium sulphate? The Magpie Trial: a randomised placebo-controlled trial. Lancet. 2002 Jun 1;359(9321):1877-90. doi: 10.1016/s0140-6736(02)08778-0. PMID 12057549
- [Background] Bergman L, Torres-Vergara P, Penny J, Wikstrom J, Nelander M, Leon J, Tolcher M, Roberts JM, Wikstrom AK, Escudero C. Investigating Maternal Brain Alterations in Preeclampsia: the Need for a Multidisciplinary Effort. Curr Hypertens Rep. 2019 Aug 2;21(9):72. doi: 10.1007/s11906-019-0977-0. PMID 31375930
- [Background] Bain ES, Middleton PF, Crowther CA. Maternal adverse effects of different antenatal magnesium sulphate regimens for improving maternal and infant outcomes: a systematic review. BMC Pregnancy Childbirth. 2013 Oct 21;13:195. doi: 10.1186/1471-2393-13-195. PMID 24139447
- [Background] Anjum S, Goel N, Sharma R, Mohsin Z, Garg N. Maternal outcomes after 12hours and 24hours of magnesium sulfate therapy for eclampsia. Int J Gynaecol Obstet. 2016 Jan;132(1):68-71. doi: 10.1016/j.ijgo.2015.06.056. Epub 2015 Oct 14. PMID 26604159
- [Background] Beyuo T, Lawrence E, Langen ES, Oppong SA. Open-labelled randomised controlled trial of 12 hours versus 24 hours modified Pritchard regimen in the management of eclampsia and pre-eclampsia in Ghana (MOPEP Study): study protocol. BMJ Open. 2019 Oct 22;9(10):e032799. doi: 10.1136/bmjopen-2019-032799. PMID 31641005
- [Background] Padda J, Khalid K, Colaco LB, Padda S, Boddeti NL, Khan AS, Cooper AC, Jean-Charles G. Efficacy of Magnesium Sulfate on Maternal Mortality in Eclampsia. Cureus. 2021 Aug 20;13(8):e17322. doi: 10.7759/cureus.17322. eCollection 2021 Aug. PMID 34567870